CLINICAL TRIAL: NCT05204459
Title: Investigating the Longitudinal Relationships Between Visual Pathway Injury, Radiological and Blood Biomarkers in Multiple Sclerosis and Related Disorders
Brief Title: MS-ResearchBiomarkerS
Acronym: MS-ReBS
Status: Recruiting | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Omar Al-Louzi, Staff Physician; Director, Visual Outcomes Lab, Cedars-Sinai Medical Center
Other Study IDs: STUDY00001690
Record Dates: First submitted 2022-01-11; First posted 2022-01-24 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive; Clinically Isolated Syndrome; Radiologically Isolated Syndrome; Neuromyelitis Optica Spectrum Disorders; Myelin Oligodendrocyte Glycoprotein Antibody-associated Disease; Neurologic Autoimmune Disease; Neurologic Disorder; Healthy Aging
Keywords: Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Primary Progressive; Multiple Sclerosis, Secondary Progressive; Clinically Isolated Syndrome; Radiologically Isolated Syndrome; Neuromyelitis Optica Spectrum Disorders; Myelin oligodendrocyte glycoprotein antibody-associated disease; Neurologic Autoimmune Disease; Neurologic Disorder; Healthy Aging
MeSH Terms: conditions — Multiple Sclerosis; Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Neuromyelitis Optica; Myelin Oligodendrocyte Glycoprotein Antibody-Associated Disease; Autoimmune Diseases of the Nervous System; Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * 2 red top tubes for serum collection (10 mL of blood each)
  * 2 purple top tube for DNA, Plasma, and Buffy Coat (10 mL of blood each)
  * 1 green top tube(10 mL of blood each)
  * 1 BD Vacutainer® CPT™ Tube with Sodium Citrate (part of an additional stem cell/genetic study blood draw; 8-10 mL of blood each)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- RRMS, SPMS, PPMS, CIS or RIS: Multiple Sclerosis (relapsing-remitting, primary or secondary progressive forms), clinically isolated syndrome, or radiologically isolated syndrome
- NMOSD: Neuromyelitis optica spectrum disorders
- MOGAD: Myelin oligodendrocyte glycoprotein antibody disorders
- Neurological disorder other than MSRD: Neurological disorders due to neurodegenerative, vascular, or headache conditions that are not related to multiple sclerosis or related disorders.
- Healthy controls: Healthy controls with no known neurological conditions

SUMMARY:
This study is being conducted to investigate risk factors for disability progression in Multiple Sclerosis and related disorders (MSRD). The primary goal is to assess whether combining information from visual assessment, blood markers, as well as historical and ongoing longitudinal MRIs of the brain, orbit (the part of the skull where eyes are located), and/or spinal cord can predict changes in quantitative disability measures related to MSRD and neurological disease.

DETAILED DESCRIPTION:
Screening:

Prospective participants will be screened at Cedars-Sinai Medical Center (CSMC) through a comprehensive review of their medical and MRI records done as part of standard of care to determine if they are eligible to participate in this study. If they never had an MRI at CSMC, they will be asked to provide records of an MRI done at another site. If the study team determines that they are eligible to continue participating, then they will move on to the main research study.

Main Research Study:

The following items will be collected as part of the main research study:

* Demographic data and medical history, including medications, family, and social history
* Complete a series of quantitative disability assessments,
* Collection of historic MRI data obtained as part of standard of care

Optional Sub-study:

Participants are not required to take part in the optional sub-study and can choose which sub-study procedures they would want to undergo. Participants can say no to the sub-study, and still remain in the main study. The optional sub-study involves undergoing one or more of the procedures below:

* Research blood draw
* Additional blood sample for a genetic and/or stem cell sub-study
* Visual assessment
* Research MRI

How long will participants be in the study? There is no prespecified end date for this study. Participants may remain in the main study as long as they are (1) willing to participate, (2) remain eligible for the study procedures, and (3) the study remains open.

Compensation for Participating Participants will be provided a voucher to cover parking expenses at Cedars-Sinai Medical Center during their participation in this research study if they undergo the optional sub-study procedures.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who meet any one of the following diagnostic criteria:

  * Diagnosis of MS, CIS,or RIS based on the 2017 revised McDonald criteria.
  * Diagnosis of NMOSD based on the 2015 revised NMOSD consensus diagnostic criteria.
  * Diagnosis of myelin oligodendrocyte glycoprotein (MOG)-related encephalomyelitis, optic neuritis, or other associated disease.
  * Diagnosis of neurological disorders other than MSRD.
  * Healthy volunteer.
* Age ≥18.
* Able to give informed consent.

Exclusion Criteria:

* Patients will be excluded from the MRI portions of the study if they have a contraindication to MRI(metallic implantsor foreign bodies, claustrophobia, MRI-incompatible pacemakers, MRI- incompatible prosthetic heart valves).
* Patients will be excluded from the MRI portions of the study if they are pregnant, but their demographic, clinical information,and disability measures may still be captured under the study.
* Patients will be excluded from the visual assessment portions of the study if they have had any recent ocular surgery (within the past two months), refractive errors of greater than or equal to ±6 diopters or other eye diseases that may affect or confound OCT/OCTA measurements (ex., age-related macular degeneration, advanced geographic atrophy, diabetic retinopathy, glaucoma).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants with the following conditions or healthy volunteers are eligible to participate in the study:
  1. Multiple sclerosis (MS), clinically isolated syndrome (CIS), or radiologically isolated syndrome (RIS)
  2. Neuromyelitis optica spectrum disorders (NMOSD)
  3. Myelin oligodendrocyte glycoprotein (MOG) antibody associated disorders (MOGAD)
  4. Neurological disorder other than MS and related disorders
  5. Healthy volunteers
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2041-11-11 (Estimated); Study Completion 2041-11-11 (Estimated)

PRIMARY OUTCOMES:
Identifying risk factors for disability progression | 10 years
  To investigate whether combining information from peripheral blood biomarkers, retinal structural, visual function, as well as historical and ongoing longitudinal MRIs (brain, cervical, and/or thoracic spinal cord) can predict quantitative disability progression risk

SECONDARY OUTCOMES:
Effect of disease modifying therapy | 10 years
  Assess the effect modification of various Food and Drug Administration(FDA)-approved disease modifying therapy on disability risk
Identify factors associated with visual disability and optic neuropathy in multiple sclerosis and related disorders | 10 years
  Using retinal structural and functional testing, this study will track longitudinal evolution of visual dysfunction and retinal injury
Identify serum, genetic, and stem cell-derived biomarkers influencing disability risks | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Omar Al-Louzi, MD, Principal Investigator — Cedars-Sinai Medical Center; Marwa Kaisey, MD, Study Director — Cedars-Sinai Medical Center; Brooke Guerrero, MD, Study Director — Cedars-Sinai Medical Center; Laura Locke, CRNP, Study Director — Cedars-Sinai Medical Center; Pascal Sati, PhD, Study Director — Cedars-Sinai Medical Center; Nancy Sicotte, MD, Study Chair — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Cedars-Sinai Clinical Research Website — https://www.cedars-sinai.org/programs/neurology-neurosurgery/clinical-trials/ms-research-biomarkers.html